CLINICAL TRIAL: NCT06853457
Title: A Transfer Learning Radiomics Model for Predicting Response to Initial Transarterial Embolization in Patients with Gastroenteropancreatic Neuroendocrine Tumor Liver Metastases: from Lesion-targeted to Patient-targeted Prediction
Brief Title: A Transfer Learning Radiomics Model for Predicting Response to Initial Transarterial Embolization in Patients with Gastroenteropancreatic Neuroendocrine Tumor Liver Metastases
Status: Completed | Type: Observational
Sponsor: First Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Xiao-Yu Yin, Professor, First Affiliated Hospital, Sun Yat-Sen University
Other Study IDs: IIT-2023-983
Record Dates: First submitted 2025-02-23; First posted 2025-03-03 (Actual); Last update posted 2025-03-03 (Actual); Status verified 2025-02

CONDITIONS: Neuroendocrine Tumors, NET
MeSH Terms: conditions — Neuroendocrine Tumors

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- training set: The training set consisted of patients from January 2014 to December 2020.
- testing set: the testing set included patients from January 2021 to September 2022.

SUMMARY:
To develop and validate a CT-based transfer learning radiomics model for predicting response to initial TAE in GEP-NETLM patients and compare its performance with traditional radiomics and clinical models.

ELIGIBILITY:
Inclusion Criteria:

* (a) Clinical diagnosed as gastroenteropancreatic neuroendocrine tumor liver metastases; (b) Received initial transarterial embolization therapy; (c) Underwent multi-phase ceCT scans pre-TAE (≤1 month) and post-TAE (4-6 weeks).

Exclusion Criteria:

* (a) Neuroendocrine carcinoma (NEC) or other malignancies. (b) Received other liver metastasis treatments. (c) Lack of Multi-phase ceCT scans records. (d) CT images with artifacts or no visible lesions.

Ages: 18 Years to 78 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study retrospectively included gastroenteropancreatic neuroendocrine tumors liver metastasis patients who receive initial transarterial embolization from January 2014 to September 2022 at The First Affiliated Hospital of Sun Yat-sen University.
Sampling Method: Probability Sample
Enrollment: 257 (Actual)
Dates: Start 2014-01-01 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2024-09-01 (Actual)

PRIMARY OUTCOMES:
The efficacy of TAE | Within one month prior and 4-6 weeks following the initial TAE.
  Complete multiphase contrast-enhanced CT images were collected preoperatively and postoperatively. The efficacy of TAE was assessed based on RECIST 1.1 criteria. Patients were classified as objective responders (those achieving complete response [CR] or partial response [PR]) or non-responders (those with stable disease [SD] or progressive disease [PD]) through evaluation of target lesions.